CLINICAL TRIAL: NCT01099631
Title: A Phase 1 Study of an IL-2 Expressing, Attenuated Salmonella Typhimurium in Patients With Unresectable Hepatic Spread From Any Non-Hematologic Primary
Brief Title: IL-2 Expressing, Attenuated Salmonella Typhimurium in Unresectable Hepatic Spread
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS003; 0906M68041 (Other: IRB, University of Minnesota); Protocol #0907-991 (Other: NIH OBA)
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Cancer of the Liver; Liver Cancer; Hepatoma; Liver Neoplasms; Biliary Cancer
Keywords: Salmonella typhimurium; unresectable hepatic cancer; attenuated Salmonella typhimurium; IL-2
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Salmonella typhimurium 10 to the 5th - Level 1 (Experimental): Patients will receive (a minimum of 3 patients) escalating doses of Salmonella typhimurium to achieve a maximum tolerated dose (MTD).
  Interventions: Biological: Salmonella typhimurium
- Salmonella typhimurium 10 to the 6th -- Level 2 (Experimental): Patients will receive (a minimum of 3 patients) escalating doses of Salmonella typhimurium to achieve a maximum tolerated dose (MTD).
  Interventions: Biological: Salmonella typhimurium
- Salmonella typhimurium 10 to the 7th -- Level 3 (Experimental): Patients will receive (a minimum of 3 patients) escalating doses of Salmonella typhimurium to achieve a maximum tolerated dose (MTD).
  Interventions: Biological: Salmonella typhimurium
- Salmonella typhimurium 10 to the 8th - Level 4 (Experimental): Patients will receive (a minimum of 3 patients) escalating doses of Salmonella typhimurium to achieve a maximum tolerated dose (MTD).
  Interventions: Biological: Salmonella typhimurium
- Salmonella typhimurium 10 to the 9th - Level 5 (Experimental): Patients will receive (a minimum of 3 patients) escalating doses of Salmonella typhimurium to achieve a maximum tolerated dose (MTD).
  Interventions: Biological: Salmonella typhimurium
- Salmonella typhimurium 10 to the 10th - Level 1 (Experimental): Patients will receive (a minimum of 3 patients) escalating doses of Salmonella typhimurium to achieve a maximum tolerated dose (MTD).
  Interventions: Biological: Salmonella typhimurium

INTERVENTIONS:
Biological: Salmonella typhimurium — Attenuated Salmonella typhimurium (virulent strain x4550) will be given orally in escalating dose groups: Level 1 = 10^5, Level 2 = 10^6, Level 3 = 10^7, Level 4 = 10^8, Level 5 = 10^9, Level 6 = 10^10.

SUMMARY:
The working hypothesis is that oral administration of an attenuated strain of Salmonella typhimurium is safe and efficacious for patients with unresectable hepatic metastasis from a solid tumor cancer. The primary objective of the study is to determine the MTD of Salmonella typhimurium in the treatment.

DETAILED DESCRIPTION:
This phase I study will be done to evaluate a dose escalation scheme of oral administration of an attenuated strain of Salmonella typhimurium expressing human interleukin-2 (IL-2) in patients with unresectable hepatic metastases from a solid tumor cancer. Standard Phase I dose escalation scheme will be used to determine the MTD of Salmonella Typhimurium. Six dose levels of Salmonella will be studied with a minimum of 3 patients enrolled in a dose level.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of malignancy (any solid tumor type) that has spread to the liver and deemed unresectable, and for which no effective standard therapies are available. Patients with additional disease outside of the liver will be allowed.
* Patients may have received any number of other prior therapies; however at least 3 weeks must have passed since last dose of chemotherapy or radiotherapy (6 weeks for Nitrosoureas or Mitomycin C) prior to study entry.
* Must have recovered from all acute toxicities (defined per National Cancer Institute's Common Toxicity Criteria for Adverse Events 3.0 ≤ grade 1) associated with previous treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy of greater than 2 months as determined by the enrolling investigator
* Adequate organ function within 1 week of treatment start defined as:

  * Adequate bone marrow reserve: leukocytes ≥ 3,000/μl, absolute neutrophil count (ANC) ≥ 1,500/μl, platelets ≥ 100,000/μl
  * Hepatic: bilirubin ≤1.5 times institutional upper limit of normal (×ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN
  * Renal: serum creatinine ≤ 1.5 x ULN
* Women of child-bearing potential and sexually active men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Unable to take oral drugs or clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: malabsorption syndrome, major resection of stomach or small bowel
* Receiving any other investigational agents
* Known central nervous system metastases
* Residing in a household or having close contact with pregnant women, young children (under the age of 1 year) or immune compromised persons
* Engaged in activities that might pose a risk for widespread dissemination of this organism, including, but not limited to; health care, child care, or food service.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations.
* Pregnant or breastfeeding. Women of child bearing potential must have a negative serum or urine pregnancy test within 7 days of prior to the start of treatment. Pregnancy testing is not required for post-menopausal or surgically sterilized women. Breast-feeding mothers will be asked to discontinue feeding infants prior to enrolling in the study.
* Known HIV infection, need for chronic steroids or other immunosuppressant drugs, or other medical conditions that in the investigator's opinion result in a significant degree of immunosuppression. Patients without identified HIV risk factors are not required to have HIV testing to be eligible.
* Known active hepatitis B or C infection
* Known HLA B27
* Have permanent artificial implants (such as, but not limited to prosthetic valves and joints.)
* Any other condition which in the investigator's opinion renders the patient at high risk for overwhelming infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W. Greeno, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Edward W. Greeno, MD, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Salmonella Typhimurium 10 to the 5 th - Level 1: Patients received Level 1 = 10^5 dose of of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 6 th - Level 2: Patients received Level 2 = 10^6th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 7 th - Level 3: Patients received Level 3 = 10^7th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 8 th - Level 4: Patients received Level 4 = 10^7th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 9th - Level 5: Patients received Level 5 = 10^9th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 10 th - Level 6: Patients received Level 6 = 10^10th dose of Salmonella typhimurium
Period: Overall Study
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6
Started | 6 | 3 | 3 | 3 | 3 | 4
Completed | 6 | 3 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Salmonella Typhimurium 10 to the 5 th - Level 1: Patients received Level 1 = 10^5th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 8 th - Level 4: Patients received Level 4 = 10^8th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 9 th - Level 5: Patients received Level 5 = 10^9th dose of Salmonella typhimurium
- Total: Total of all reporting groups
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9 th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6 | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 4 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 1 | 0 | 3 | 12
  >=65 years | 2 | 1 | 1 | 2 | 3 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 1 | 2 | 2 | 11
  Male | 2 | 2 | 2 | 2 | 1 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 3 | 3 | 3 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 1 | 0 | 3
  White | 6 | 1 | 3 | 3 | 1 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Events to Determine the Maximum Tolerated Dose (MTD) of Salmonella Typhimurium
Description: Maximum tolerated dose will be determined by the number of patients with Dose limiting toxicity (DLT) at a given dose level. DLT is defined as treatment related: Sepsis (salmonella) syndrome, Grade 4 vomiting or diarrhea, Other grade 3 or greater toxicity. If > or = 2 patients at a dose level has a DLT, this level will be declared the MTD.
Time Frame: Up to 24 Weeks After Dose of Salmonella typhimurium
Measure: Count of Participants; unit: Participants
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Complete Response to Treatment
Description: Evaluation is performed using Response Evaluation Criteria in Solid Tumors (RECIST). Each patient will be assigned one of the following categories: Complete response (CR) the disappearance of all target lesion; Partial response (PR) at least a 30% decrease; Progressive disease (PD) at least a 20% increase, or the appearance of one or more new lesions; Stable disease (SD) neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease; early death from malignant disease; unknown (insufficient evaluation to determine response status).
Time Frame: 8 Weeks After Treatment with Salmonella Typhimurium
Measure: Count of Participants; unit: Participants
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Peripheral Blood NK Cells Count
Description: Patients receiving doses of 10^5 through 10^10 Colony forming units of Salmonella typhimurium had their peripheral blood flow cytometry performed to identify the NK (Natural killer) cells population (CD8-, CD4-, CD49b+) prior to administration and at 5 weeks post administration.
  The flow cytometry data below was gathered by gating on the lymphocyte population of cells in the patient's blood, as determined by FSC vs. SSC. The mean percentage of NK cells in sample's lymphocyte population is given.
Time Frame: Baseline and 5 Weeks After Dosing with Salmonella typhimurium
Population: One patient in 10 to the 6 th - Level 2 arm was not evaluable. One patient in 10 to the 7 th - Level 3 arm was not evaluable. Two patients in 10 to the 8 th - Level 4 arm were not evaluable. Two patients in 10 to the 9th - Level 5 arm were not evaluable. Two patients in 10 to the 10th - Level 6 arm were not evaluable.
Measure: Mean (Standard Deviation); unit: peripheral NK cells percentage
Groups:
- Salmonella Typhimurium 10 to the 8 th - Level 4: Patients received Level 4 = 10^8 th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 10 th - Level 6: Patients received Level 1 = 10^10 th dose of Salmonella typhimurium
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6
Number analyzed (Participants) | 6 | 2 | 2 | 1 | 1 | 2
peripheral NK cells percentage
  Before administration | 10.52 (5.41) | 8.2 (2.55) | 17.1 (3.3) | 23.5 (0) | 19.6 (0) | 6.55 (0.49)
  After administration | 13.75 (5.18) | 9.3 (3.54) | 19.7 (8.06) | 28.8 (0) | 23.9 (0) | 5.65 (0.91)

4. Secondary Outcome: Peripheral Blood T Cells Count
Description: Patients receiving doses of 10^5 through 10^10 Colony forming units of Salmonella typhimurium had their peripheral blood flow cytometry performed to identify the NK (Natural killer) cells population (CD25+, FoxP3+) prior to administration and at 5 weeks post administration.
  The flow cytometry data below was gathered by gating on the lymphocyte population of cells in the patient's blood, as determined by FSC vs. SSC. The mean percentage of T cells in sample's lymphocyte population is given.
Time Frame: Baseline and 5 Weeks After Dosing with Salmonella typhimurium
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent peripheral blood T cells
Groups:
- Salmonella Typhimurium 10 to the 6 th - Level 2: Patients received Level 2 = 10^6 th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 7 th - Level 3: Patients received Level 3 = 10^7 th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 9th - Level 5: Patients received Level 5 = 10^10 th dose of Salmonella typhimurium
- Salmonella Typhimurium 10 to the 10 th - Level 6: Patients received Level 6 = 10^10 th dose of Salmonella typhimurium
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6
Number analyzed (Participants) | 6 | 2 | 2 | 1 | 1 | 4
percent peripheral blood T cells
  Before administration | 51.77 (20.04) | 50.25 (8.70) | 63 (2.82) | 56.3 (0) | 50.1 (0) | 70.6 (7.35)
  After administration | 53.92 (9.17) | 64.25 (8.98) | 45.3 (20.85) | 42.4 (0) | 53.2 (0) | 77.65 (1.63)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Salmonella Typhimurium 10 to the 5 th - Level 1 | Salmonella Typhimurium 10 to the 6 th - Level 2 | Salmonella Typhimurium 10 to the 7 th - Level 3 | Salmonella Typhimurium 10 to the 8 th - Level 4 | Salmonella Typhimurium 10 to the 9 th - Level 5 | Salmonella Typhimurium 10 to the 10 th - Level 6
All-Cause Mortality (participants affected / at risk) | 4/6 | 2/3 | 3/3 | 3/3 | 2/3 | 4/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 3/3 | 3/3 | 2/3 | 1/4
Other Adverse Events (participants affected / at risk) | 4/6 | 2/3 | 3/3 | 3/3 | 2/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salmonella Typhimurium 10 to the 5 th - Level 1 (N=6) | Salmonella Typhimurium 10 to the 6 th - Level 2 (N=3) | Salmonella Typhimurium 10 to the 7 th - Level 3 (N=3) | Salmonella Typhimurium 10 to the 8 th - Level 4 (N=3) | Salmonella Typhimurium 10 to the 9 th - Level 5 (N=3) | Salmonella Typhimurium 10 to the 10 th - Level 6 (N=4)
New compression fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
GI bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hyperkalemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salmonella Typhimurium 10 to the 5 th - Level 1 (N=6) | Salmonella Typhimurium 10 to the 6 th - Level 2 (N=3) | Salmonella Typhimurium 10 to the 7 th - Level 3 (N=3) | Salmonella Typhimurium 10 to the 8 th - Level 4 (N=3) | Salmonella Typhimurium 10 to the 9 th - Level 5 (N=3) | Salmonella Typhimurium 10 to the 10 th - Level 6 (N=4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 1 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Fever (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (3)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes